CLINICAL TRIAL: NCT04411342
Title: Prevalence of Normoalbuminuric Chronic Kidney Disease and Its Risk Factors in Patients With Type 2 Diabetes Attending the Diabetes Center of Assiut University Hospital
Brief Title: Normoalbuminuric Chronic Kidney Disease in Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Michael Wadae, clinical investigator, Assiut University
Other Study IDs: normoalbuminuric CKD in DM2
Record Dates: First submitted 2020-03-12; First posted 2020-06-02 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with type 2 diabetes: patients with type 2 diabetes and have normal range of albumine in urine and decline in renal functions
  Interventions: Diagnostic Test: Albumin creatinine ratio

INTERVENTIONS:
Diagnostic Test: Albumin creatinine ratio — normal range of albumin in urine in patients with type 2 diabetes

SUMMARY:
* Assess the prevalence of normoalbuminuric CKD in Type 2 diabetes.
* Study the risk factors of normoalbuminuric CKD in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is considered a major cause of chronic kidney disease (CKD), where about 40% of the diabetics develop diabetic kidney disease (DKD) resulting in albuminuria, reduction of glomerular filtration rate (GFR), or both .

Albuminuria was widely considered the first clinical sign of DKD, therefore, it has been used as a screening test for DKD. However, recent studies showed that a significant number of T2DM patients have a decreased GFR with normoalbuminuria, known as non-albuminuric DKD (NA-DKD) .

The use of albuminuria as an early marker of DKD onset or progression requires a careful interpretation because in diabetics, albuminuria has a great tendency to return to normal spontaneously. Evidence based studies reported that about 18-51 percent of T2DM (followed during 2-10 years) present first with albuminuria turn to normoalbuminurics spontaneously during the period of follow-up .

The United Kingdom Prospective Diabetes Study (UKPDS) reported that some diabetics pass directly from a normoalbuminuria to renal insufficiency (0.1% per year) .

Albuminuria as a marker of glomerular lesion progression has some limitations because of its intra-patient variability and possibility of spontaneous regress (in >50% of the patients with low levels of albuminuria), in contrast with GFR that has low variability and infrequent improvement .

Few of T2DM patients are presented without significant proteinuria but present with renal insufficiency and developed DKD (i.e., estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2), which was defined as normoalbuminuric diabetic kidney disease (NADKD) or diabetic kidney disease without proteinuria where albuminuria does not associate with impairment of kidney function .

The ADA criteria for diagnosis of DKD now involve the presence of eGFR < 60 mL/min/1.73 m2 or the presence of UAE > 30 mg/24 h. In patients with NADKD, the risk factors include obesity, hypertension, high TG levels, sex, smoking, poor glycemic control, and glomerular hyperfiltration which play a role in nephrosclerosis. Macroangiopathy is also prevalent in patients with NADKD .

Intrarenal arteriosclerosis is the main cause of renal impairment in type 2 diabetic patients independent of albuminuria, and this partly cause eGFR decline in these patients. Several studies also suggest that decline in renal function is mainly due to interstitial injury (a pathological change in DN) as compared with glomerular injury .

Normoalbuminuria is associated with Diabetic kidney disease (DKD), which is the commonest cause of end-stage renal disease (ESRD) all over the world. The clinical manifestations of DKD consist of a progressive increase in albuminuria and a decline in estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2. Hence, the diagnosis of DKD in patients with declining renal function without albuminuria is more difficult. The decline of renal function is slower in normoalbuminuria .

Tthe majority of patients with DKD had albuminuria, but a significant proportion had the normoalbuminuric renal impairment (46.6%) . The prevalence of NADKD ranges globally from 14.29 to 56.6% among diabetic patients with different ethnicities .

The prevalence of NADKD is about 23.3% to 56.6% in T2DM patients with a decline in the renal function presented with normal albuminuria . However, the prevalence at which the patients develop normoalbuminuric renal impairment in Type 2 diabetes are not completely defined.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 -65 years .
* Diagnosed previously with T2DM.

Exclusion Criteria:

* Patients with type 1 diabetes,

  * Patients with secondary diabetes,
  * Patients with gestational diabetes
  * Patients with severe acute or chronic hepatic or cardiac diseases.
  * Patients with Past or present history of malignancy .
  * Patients with in need for renal replacement therapy.
  * Patients with other probable causes for CKD.
  * Patients with an active urinary sediment and nephrotic - range proteinuria .

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with type 2 diabetes attending diadetes center of Assiut University
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Normoalbuminuric chronic kidney disease | Baseline
  The required sample size(200 patients) has been calculated using the EPI info version which achieve power of study 80%.

IPD SHARING:
Plan to Share IPD: No